CLINICAL TRIAL: NCT03958422
Title: A Randomized, Single-blind, Controlled Clinical Trial of Cardiomyopeptidin Intervention in Patients With Acute ST-segment Elevation Myocardial Infarction Undergoing Direct PCI After Ischemia-reperfusion Injury
Brief Title: Clinical Study of Cardiomyopeptidin on Postoperative Ischemia-reperfusion Injury in Patients With Primary PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dalian Zhen-Ao Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLZA2019P01
Record Dates: First submitted 2019-04-18; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-04

CONDITIONS: Survival Myocardial Area After Acute Myocardial Death; Left Ventricular Ejection Fraction
Keywords: Acute myocardial infarction; Nuclear magnetic image; Survival myocardial area
MeSH Terms: interventions — cardiomyopeptidin

STUDY DESIGN:
Intervention Model Description: Random, controlled, single blind
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myocardin test group (Experimental): Patients in cardiomyopeptidin group are given the injection of cardiomyopeptidinl before primary percutaneous coronary intervention (PCI) and intravenous infusion of cardiomyopeptidin was performed 3 days after primary PCI.
  Interventions: Drug: cardiomyopeptidin
- Blank test group (No Intervention): Patients in blank test group aren't given the injection of cardiomyopeptidinl before primary percutaneous coronary intervention (PCI) .

INTERVENTIONS:
Drug: cardiomyopeptidin — The main component of cardiomyopeptidin is the peptide active substance extracted from the ventricular myocytes of healthy young pigs.
  Arms: Myocardin test group

SUMMARY:
In this study, advanced techniques of myocardial nuclear magnetic perfusion scanning were used to quantitatively assess infarct size after acute myocardial infarction, saved viable myocardium, and microcirculatory obstruction area. Objectively and quantitatively evaluate early use of cardiomyopeptidin for direct PCI of ST-segment elevation myocardial infarction. After the improvement of microcirculation and increase the intervention effect of viable myocardium.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, single-blind, single-center clinical trial. Patients with ST-segment elevation myocardial infarction (STEMI) who were admitted in the People's Liberation Army General Hospital were equally randomized to receive either cardiomyopeptidin or placebo, and patients in cardiomyopeptidin group are given the injection of cardiomyopeptidinl before primary percutaneous coronary intervention (PCI) and intravenous infusion of cardiomyopeptidin was performed 3 days after primary PCI. Myocardial perfusion flow grade was evaluated by the result of primary PCI. Myocardial infarct size, microvascular obstruction and salvage myocardium were evaluated by enhanced cardiac magnetic resonance (CMR). Major adverse cardiovascular events (nonfatal myocardial infarction, all-cause death, hospitalization for acute heart failure, and revascularization for angina) were observed during the 6-month follow-up. CMR is performed to evaluate the effect of cardiomyopeptidin before primary PCI on myocardial salvage and microcirculation perfusion in patients with STEMI.

ELIGIBILITY:
Inclusion Criteria:

* 1) Sign the informed consent form;
* 2) Age ≥ 18 and ≤ 80 years old, gender is not limited;
* 3) Defining the diagnosis of acute myocardial infarction, with indications for direct coronary intervention;
* 4) Ischemic chest pain lasts for more than 30 minutes and adjacent ST or 2 leads of more than 2 or more leads (limb lead ≥ 0.1 mV, chest lead ≥ 0.2 mV) with or without elevated myocardial enzyme levels ;
* 5) The course of disease is ≤12 hours or accompanied by cardiogenic shock or heart failure (onset >12h).

Exclusion Criteria:

* (1) Cardiogenic shock, Killip III-IV grade, papillary muscle rupture, interventricular septal perforation, ventricular ventricular fibrillation and electrical cardioversion, and III degree AVB implantation of temporary pacemaker before PCI;
* (2) LVEF ≤ 30%;
* (3) Previous history of PCI and CABG history;
* (4) acute and chronic infectious diseases (severe pneumonia, etc.);
* (5) Recent history of hemorrhagic stroke (within six months);
* (6) Combining liver and kidney dysfunction caused by various reasons;
* (7) History of valvular heart disease;
* (8) Congenital heart disease and pulmonary hypertension;
* (9) History of various types of cardiomyopathy;
* (10) bleeding and other thrombotic diseases;
* (11) severe anemia, thrombocytopenia and other blood system diseases;
* (12) Patients with malignant tumors, autoimmune diseases, and various causes of glucocorticoids and immunosuppressive agents;
* (13) Patients with a history of drug allergy, allergic diseases or allergies, or patients who are allergic to any of the ingredients in this product;
* (14) Patients with severe mental or neurological diseases;
* (15) pregnant women, lactating women, and subjects with a pregnancy plan during the trial;
* (16) According to the investigator's judgment, the subject is unable to complete the study or may not be able to comply (for administrative reasons or other reasons) the subjects required for this study.
* (17) Patients who have participated in other clinical trials in the past 3 months.Researchers believe that it is not appropriate to participate in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarct size | 7±3 days after surgery
  Nuclear magnetic imaging focused on the assessment of myocardial infarct size（%）;

SECONDARY OUTCOMES:
Delay enhancement | 7±3 days after surgery
  Nuclear magnetic imaging focused on microcirculation obstruction, myocardial edema area, delayed enhancement
ECG ST-T changes | "hour6", "hour12","hour24"after myocardial infarction
  Interpretation of ST-T changes in leads based on electrocardiogram
Heart function classification | "day6", "week4","week12","week24"after surgery
  Cardiac function grading of patients with acute myocardial infarction by Killip grading
CK（ng/ml） | "hour6", "hour12","hour24" and 7±3 days after myocardial infarction
  one of Myocardial enzymes CK-MB(ng/ml)、cTnT(ng/ml)、BNP(pg/ml)
CK-MB(ng/ml) | "hour6", "hour12","hour24" and 7±3 days after myocardial infarction
  one of Myocardial enzymes cTnT(ng/ml)、BNP(pg/ml)
cTnT(ng/ml) | "hour6", "hour12","hour24" and 7±3 days after myocardial infarction
  one of Myocardial enzymes
BNP(pg/ml) | "hour6", "hour12","hour24" and 7±3 days after myocardial infarction
  one of Myocardial enzymes
Cardiac echocardiography | 3days and 1,3,6 monthes after myocardial infarction
  Left ventricular ejection fraction
Incidence of cardiovascular events | 7±3 days and 1,3,6 monthes after myocardial infarction
  Non-lethal myocardial infarction, all-cause death, revascularization due to angina pectoris, re-hospitalization of acute heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Study Director — cardiology

IPD SHARING:
Plan to Share IPD: Undecided